CLINICAL TRIAL: NCT04732923
Title: Maintenance of Physical Condition and Physical Activity at One Year After Cardiac Rehabilitation Program
Acronym: APA&Co
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Cholet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC_2020_0001
Record Dates: First submitted 2021-01-15; First posted 2021-02-01 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-04

CONDITIONS: Coronary Disease; Acute Coronary Syndrome
Keywords: physical condition; physical activity; cardiac rehabilitation
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): This study is defined in 3 stages :
  STEP 1 : during the cardiac rehabilitation program over 4 weeks
  STEP 2 : monitoring at 6 months after cardiac rehabilitation program
  STEP 3 : monitoring at one year after cardiac rehabilitation program
  Interventions: Other: Assigned intervention - procedure

INTERVENTIONS:
Other: Assigned intervention - procedure — This study is defined in 3 stages :
  STEP 1 : during the cardiac rehabilitation program over 4 weeks 6 minute walk test, questionnaires
  STEP 2 : monitoring at 6 months after cardiac rehabilitation program Nurse interview, 6 minute walk test, questionnaires
  STEP 3 : monitoring at one year after cardiac rehabilitation program Nurse interview, 6 minute walk test, questionnaires

SUMMARY:
Maintaining physical activity post-cardiac rehabilitation (CR) has a major role in disease progression and patient prognosis, especially given its potential impact on physical condition. Unfortunately, during a nursing interview carried out 6 months after the CR at the Center Hospitalier de Cholet, we find that 40% do not maintain regular physical activity. This observation is in line with the literature since it emerges respectively at 2 months and 1 year post-CR that between 47% and 59% of patients do not comply with the recommendations in terms of physical activity (Guiraud et al, 2012).

However, data suggest that during the post-CR follow-up phase at 6 months, there could be a maintenance of the physical condition assessed via the distance at the 6-minutes walk test (Pavy et al, 2012; Racodon et al, 2019). There is a lack of data on the maintenance of physical condition beyond 6 months since no study has evaluated the maintenance of physical condition at 1 year post-CR by 6-minutes walk test.

DETAILED DESCRIPTION:
The objective of this study is to examine the maintenance of physical condition at one year after cardiac rehabilitation program by the 6-minutes walk test.

ELIGIBILITY:
Inclusion Criteria :

* Patient participating in cardiac rehabilitation
* Patient who presented an acute coronary syndrome
* Patient having signed the written consent to participate
* Patient able to comply with the constraints of the protocol

Exclusion Criteria :

* Patient with heart failure
* Patient reluctant or unable to comply with the protocol
* Pregnant, parturient and nursing mothers
* Persons deprived of their liberty or under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
to study the maintenance of physical condition after cardiac rehabilitation program | at one year
  6-minutes walk test

SECONDARY OUTCOMES:
to study the maintenance of physical condition after cardiac rehabilitation program | at 6 months
  6-minutes walk test
to study physical activity during the monitoring | at 6 months and one year
  questionnaire IPAQ
to study the motivation for physical activity during the monitoring | at 6 months and one year
  questionnaire EMAPS
to study obstacles to maintaining physical activity | at one year
  nurse interview

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vollot, Study Director — Centre Hospitalier de Cholet; Paul Da Ros Vettoretto, Principal Investigator — Centre Hospitalier de Cholet
Locations (1):
- Centre Hospitalier de CHOLET, Cholet, France

IPD SHARING:
Plan to Share IPD: No